CLINICAL TRIAL: NCT05608018
Title: A Novel Distracted Driving Prevention Technology Phase II
Brief Title: Preventing Distracted Driving Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnesota HealthSolutions (Industry)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21-018977
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Distracted Driving
Keywords: mobile phone use while driving

STUDY DESIGN:
Intervention Model Description: This study is a randomized control trial with 2 arms, and 4 possible randomization groups (intervention/Bluetooth, intervention/non-Bluetooth, control/Bluetooth, and control/non-Bluetooth). The control group will receive the control condition, during which the app monitors driving but the intervention feature is not enabled, and the intervention group will receive the intervention condition during which the intervention feature is enabled. Both groups will self-report their smartphone communication while driving via periodic surveys. Participants randomized to receive a Bluetooth device will keep the device in their primary vehicle for the duration of the study. This device will collect outgoing text date and time from their dyad partner enrolled in the study. Non-Bluetooth participants will not receive the device.
Who Masked: Participant
Masking Description: Participants will be randomly assigned to the intervention/Bluetooth group, intervention/non-Bluetooth group, control/Bluetooth group, or control/non-Bluetooth group upon enrollment in the study. Assignment status will not be concealed from the research assistants enrolling the participant, the participants themselves, or the rest of the study team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Bluetooth (Other): Participants receive a the same app as the intervention group, but the feature that notifies the teens parent when they are driving is turned off. They will self-report their smartphone communication while driving via periodic surveys. Participants will receive a Bluetooth device to keep in their primary vehicle for the duration of the study.
  Interventions: Other: Control Bluetooth
- Intervention Bluetooth (Other): Participant received the app with all features turned on, so the parent gets a notification when the teen is driving before they go to send a text message to the teen. They will self-report their smartphone communication while driving via periodic surveys. Participants will receive a Bluetooth device to keep in their primary vehicle for the duration of the study.
  Interventions: Other: Intervention Bluetooth
- Control non-Bluetooth (Other): Participants receive a the same app as the intervention group, but the feature that notifies the teens parent when they are driving is turned off. They will self-report their smartphone communication while driving via periodic surveys. Participants will not receive a Bluetooth device.
  Interventions: Other: Control non-Bluetooth
- Intervention non-Bluetooth (Other): Participant received the app with all features turned on, so the parent gets a notification when the teen is driving before they go to send a text message to the teen. They will self-report their smartphone communication while driving via periodic surveys. Participants will not receive a Bluetooth device.
  Interventions: Other: Intervention non-Bluetooth

INTERVENTIONS:
Other: Intervention Bluetooth — Participants will receive a Bluetooth device to use for the duration of the study, and will use the app with all features turned on.
  Arms: Intervention Bluetooth
Other: Intervention non-Bluetooth — Participants will not receive a Bluetooth device, and will use the app with all features turned on.
  Arms: Intervention non-Bluetooth
Other: Control Bluetooth — Participants will receive a Bluetooth device to use for the duration of the study, and will use the app with some features turned off.
  Arms: Control Bluetooth
Other: Control non-Bluetooth — Participants will not receive a Bluetooth device, and will use the app with some features turned off.
  Arms: Control non-Bluetooth

SUMMARY:
The purpose of the study is to determine the efficacy of a smartphone app in reducing mobile phone use while driving among teens and parents. Prior to sending a message, the smartphone app informs a potential message sender that the recipient is driving.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether the app reduces (1) smartphone communication sent from parent to teen while the teen is driving; and (2) smartphone communication sent from teen while the teen is driving. The secondary objectives are to: Determine whether the app reduces smartphone communication sent from teen to parent while parent is driving; Evaluate the acceptability of the app among parents and teens; and determine the relationship between individual differences (demographics, typical smartphone use, driving history, risk perception) and the app's efficacy.

ELIGIBILITY:
Inclusion Criteria:

Teen participants:

1. 16 to 19 years of age
2. Hold a valid driver's license
3. Own an iPhone
4. Drive at least 3 days per week

Parent/caregiver participants:

1. 18 to 75 years of age
2. Hold a valid driver's license
3. Own an iPhone
4. Drive at least 3 days per week

Exclusion Criteria:

Teen participants:

1. Non-fluency in written or spoken English

Parent/caregiver participants:

1. Non-fluency in written or spoken English

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Changes in frequency of smartphone use while driving | 3 weeks
  Changes in smartphone communication sent from parent to teen while the teen is driving and changes in smartphone communication sent from teen while the teen is driving. Frequency of smartphone use is recorded by the app among the three app modes. Within-driver smartphone use over the 3-week study period is compared as the app modes change. Smartphone use between driver groups will also be compared.

SECONDARY OUTCOMES:
Changes in frequency of self-reported smartphone use while driving | 3 weeks
  The change in self-reported smartphone use while driving will be assessed using the same within-driver and between-driver comparisons as the primary outcome measure. Self-reported smartphone use is collected through 10 items on a participant survey that is completed at enrollment, each week for 3 weeks. Participants also report how many times per day (free text, any number greater than or equal to 0) that they drove, and talked on a hands-held smartphone, sent a text, and read a text while driving.
Acceptability and Usability of the App | 3 weeks
  Participant assessment of accessibility and usability will be collected, and Manual Mode and Auto-Detect Mode of the LifeSaver app will be compared. Participants complete a survey at the end of week 3, post-intervention. 8 items in the survey ask participants about accessibility and usability of the app through Likert scales (range from Not at all to Extremely). 3 items in the survey ask participants about accessibility and usability of the app through open-ended questions, where participants are able to enter free text. There is no overall score for these survey items.
Changes in frequency of text messages sent to Bluetooth device users | 3 weeks
  Bluetooth device users will have received text message date and time collected via the Bluetooth device. This device will only collect data from the dyad partner enrolled in the study with them. This data will be used to validate the self report data collected from all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Seifert, MPH, Principal Investigator — Study Principal Investigator
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and study documents will be shared with Minnesota HealthSolutions (the sponsor). No identifiable data will be used for future study without first obtaining Institutional Review Board (IRB) approval. The investigator will obtain a data use agreement between the provider (the PI) of the data and any recipient researchers (including others at CHOP) before sharing a limited dataset (PHI limited to dates and zip codes).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study will comply with CHOP's data retention policy (A-3-9). All study data will be maintained for at least 6 years following study completion. There is no set timeline for the destruction of the study's de-identified data
Access Criteria: IRB approval, data use agreement

REFERENCES:
- [Background] Durbin DR, Curry AE, García-España JF, et al. Miles to Go: Monitoring Progress in Teen Driver Safety. The Children's Hospital of Philadelphia Research Institute and State Farm Insurance Companies; 2012. http://www.teendriversource.org/tools/support_gov/detail/205.
- [Background] Curry AE, Hafetz J, Kallan MJ, Winston FK, Durbin DR. Prevalence of teen driver errors leading to serious motor vehicle crashes. Accid Anal Prev. 2011 Jul;43(4):1285-90. doi: 10.1016/j.aap.2010.10.019. Epub 2010 Nov 19. PMID 21545856
- [Background] Redelmeier DA, Tibshirani RJ. Association between cellular-telephone calls and motor vehicle collisions. N Engl J Med. 1997 Feb 13;336(7):453-8. doi: 10.1056/NEJM199702133360701. PMID 9017937
- [Background] National Highway Traffic Safety Administration. Research Note: Distracted Driving 2015. Washington, DC; 2017. https://crashstats.nhtsa.dot.gov/Api/Public/ViewPublication/812381.
- [Background] Ehsani J, Li K, Simons-Morton BG. Teenage Drivers Portable Electronic Device Use While Driving. In: ; 2015:219-225. doi:10.17077/drivingassessment.1575
- [Background] Insurance Institute for Highway Safety, Highway Loss Data Institute. Fatality Facts 2017: Teenagers. Insurance Institute for Highway Safety (IIHS). https://www.iihs.org/topics/fatality-statistics/detail/teenagers. Published 2018. Accessed August 12, 2019.
- [Background] How Teens Use Media: A Nielsen Report on the Myths and Realities of Teen Media Trends.; 2009. http://blog.nielsen.com/nielsenwire/reports/nielsen_howteensusemedia_june09.pdf.
- [Background] Pradhan AK, Hammel KR, DeRamus R, Pollatsek A, Noyce DA, Fisher DL. Using eye movements to evaluate effects of driver age on risk perception in a driving simulator. Hum Factors. 2005 Winter;47(4):840-52. doi: 10.1518/001872005775570961. PMID 16553070
- [Background] Hafetz JS, Jacobsohn LS, Garcia-Espana JF, Curry AE, Winston FK. Adolescent drivers' perceptions of the advantages and disadvantages of abstention from in-vehicle cell phone use. Accid Anal Prev. 2010 Nov;42(6):1570-6. doi: 10.1016/j.aap.2010.03.015. Epub 2010 Jul 2. PMID 20728605
- [Background] LaVoie N, Lee YC, Parker J. Preliminary research developing a theory of cell phone distraction and social relationships. Accid Anal Prev. 2016 Jan;86:155-60. doi: 10.1016/j.aap.2015.10.023. Epub 2015 Nov 10. PMID 26562672
- [Background] McDonald CC, Sommers MS. Teen Drivers' Perceptions of Inattention and Cell Phone Use While Driving. Traffic Inj Prev. 2015;16 Suppl 2(0):S52-8. doi: 10.1080/15389588.2015.1062886. PMID 26436243